CLINICAL TRIAL: NCT04220632
Title: An Open Label, Multicenter, Phase I/II Study of IBI377 in Combination With Corticosteroids for the Treatment of First-Line Acute Graft-Versus-Host Disease
Brief Title: A Study of IBI377 in Combination With Corticosteroids for the Treatment of First-Line Acute Graft-Versus-Host Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Adverse events of the first patient
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI377A201
Record Dates: First submitted 2020-01-04; First posted 2020-01-07 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: GVHD,Acute
MeSH Terms: interventions — itacitinib; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Itacitinib+corticosteroids (Experimental): Itacitinib administered in combination with corticosteroids
  Interventions: Drug: Itacitinib; Drug: Prednisone; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Itacitinib — at the protocol-defined dose administered orally once daily (QD) plus corticosteroids.
  Other Names: IBI377
Drug: Prednisone — Oral prednisone may be used to begin standard corticosteroid background treatment at the investigator's discretion, at a dose equivalent to methylprednisolone 2 mg/kg per day.
Drug: Methylprednisolone — Oral prednisone may be used to begin standard corticosteroid background treatment at the investigator's discretion, at a dose equivalent to methylprednisolone 2 mg/kg per day.

SUMMARY:
The purpose of this study is to evaluate itacitinib in combination with corticosteroids as first-line treatment of participants with Grade II to IV acute graft-versus-host disease (aGVHD).

DETAILED DESCRIPTION:
This is an open label, single-arm, multicenter Phase I/II study of IBI377 in combination with corticosteroids as first-line treatment of subjects with Grade II to IV aGVHD. In Phase I, the PK, safety, tolerability and efficacy of IBI377 will be assessed in 12 subjects. In Phase II, the efficacy and safety will be assessed in 48 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone 1 allo-HSCT(hematopoietic stem cell transplantation) from any donor (related or unrelated with any degree of HLA(human leukocyte antigen) matching) and any donor source (bone marrow, peripheral blood stem cells, or cord blood) for a hematologic malignancy or disorder. Recipients of myeloablative and reduced-intensity conditioning regimens are eligible.
* Clinically suspected Grade II to IV aGVHD as per MAGIC criteria, occurring after allo-HSCT and any GVHD prophylaxis regimen.
* Evidence of myeloid engraftment. Use of growth factor supplementation is allowed.
* Serum creatinine ≤ 2.0 mg/dL or creatinine clearance ≥ 40 mL/min measured or calculated by Cockroft Gault equation.
* Willing to avoid pregnancy or fathering children.
* Able to give written informed consent and comply with all study visits and procedures.
* Able to swallow and retain oral medication.

Exclusion Criteria:

* Has received more than 1 allo-HSCT.
* Has received more than 2 days of systemic corticosteroids for acute-GVHD.
* Presence of GVHD overlap syndrome.
* Presence of an active uncontrolled infection.
* Known human immunodeficiency virus infection.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection that requires treatment or at risk for HBV reactivation.
* Participants with evidence of relapsed primary disease, or participants who have been treated for relapse after the allo-HSCT was performed.
* Any corticosteroid therapy for indications other than GVHD at doses > 1 mg/kg per day methylprednisolone (or prednisone equivalent) within 7 days of randomization.
* Severe organ dysfunction unrelated to underlying GVHD, including.
* Cholestatic disorders or unresolved veno-occlusive disease of the liver.
* Clinically significant or uncontrolled cardiac disease.
* Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.
* Currently breast feeding.
* Received JAK(Janus kinase) inhibitor therapy after allo-HSCT for any indication. Treatment with a JAK inhibitor before allo-HSCT is permitted.
* Treatment with any other investigational agent, device, or procedure within 21 days (or 5 half-lives, whichever is greater) of enrollment.
* Any medical complications or conditions that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate based on Center for International Bloe index | 28 days
  Defined as the percentage of participants demonstrating a complete response (CR), very good partial responseod and Marrow Transplant Research (CIBMTR) respons (VGPR), or partial response (PR).

SECONDARY OUTCOMES:
Nonrelapse mortality | Month 6
  Defined as the percentage of participants who died due to causes other than malignancy relapse
Duration of response | Baseline through 30-35 days after end of treatment, expected to average approximately 6 months
  Defined as the interval from first response until GVHD progression or death.
Cmax of itacitinib when administered in combination with corticosteroids | Protocol-defined timepoints up to Day 28
  Defined as maximum observed plasma concentration.
Cmin of itacitinib when administered in combination with corticosteroids | Protocol-defined timepoints up to Day 28
  Defined as minimum observed plasma concentration
Tmax of itacitinib when administered in combination with corticosteroids | Protocol-defined timepoints up to Day 28
  Defined as time to maximum plasma concentration
AUC(area under curve) of itacitinib when administered in combination with corticosteroids | Protocol-defined timepoints up to Day 28
  Protocol-defined timepoints up to Day 28
CL/F(clearance) of itacitinib when administered in combination with corticosteroids | Protocol-defined timepoints up to Day 28
  Defined as oral dose clearance

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China